CLINICAL TRIAL: NCT01703520
Title: Finasteride and Male Breast Cancer - A Register-Based Nested Case-Control Study in Denmark, Finland, Norway, and Sweden
Brief Title: Finasteride (MK-0906) and Male Breast Cancer - A Register-Based Nested Case-Control Study (MK-0906-162/2003.021).
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Collaborators: Institute for Applied Economics and Health Research Aps (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0906-162; 2003.021 (Other: Merck)
Record Dates: First submitted 2012-09-24; First posted 2012-10-10 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Male Breast Cancer
Keywords: Males breast cancer; Finasteride; PROSCAR®; PROPECIA®
MeSH Terms: conditions — Breast Neoplasms, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Male Finasteride Users: Male finasteride users aged 35 years and above in the registries of Denmark (1995-2013), Finland (1994-2013), Norway (2008-2013), and Sweden (2005-2013).
- Male Finasteride Non-users: Country-matched male finasteride non-users aged 35 years and above in the registries of Denmark (1995-2013), Finland (1994-2013), Norway (2008-2013), and Sweden (2005-2013).
- Men with Breast Cancer: Breast cancer cases among men aged 35 years and above in the registries of Denmark (1995-2013), Finland (1994-2013), Norway (2008-2013), and Sweden (2005-2013).
- Men without Breast Cancer: Country- and age-matched controls: men without breast cancer aged 35 years and above in the registries of Denmark (1995-2013), Finland (1994-2013), Norway (2008-2013), and Sweden (2005-2013).

SUMMARY:
The objective of this study is to investigate the potential association between finasteride (MK-0906) exposure and the development of breast cancer in men residing in Denmark, Sweden, Finland, and Norway from data in national registries. The primary hypothesis of this study is that the previously reported increased incidence of male breast cancer among finasteride users is explained by confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Participant's study medical information available in population-based health and medical registries, prescription registries, and mortality registries in Denmark, Finland, Norway, or Sweden within the observation period of 1995 to 2013
* Male with breast cancer with medical information in one of the 4 country-specific registries in this study OR country- and age-matched control men without breast cancer and with medical information in one of the 4 country-specific registries
* Study participant's exposure to finasteride is available

Exclusion Criteria:

For country- and age-matched control men without breast cancer

* Previous cancer diagnosis or treatment for cancer except non-melanoma skin cancer
* Previous prostatectomy
* Finasteride or dutasteride use (dutasteride is a drug in the same class as finasteride) within first 6 months of registration in the prescription registers (new user design).

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population-based health and medical registries, prescription registries, and mortality registries in Denmark, Finland, Norway, and Sweden
Sampling Method: Probability Sample
Enrollment: 575216 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Stage 1 - Person-Years of Exposure to Finasteride by Participant Age and Year | Up to 14 years
Stage 1 - Initial Incidence Rates of Male Breast Cancer Stratified by Exposure to Finasteride | Up to 14 years
Stage 1 - All-Cause Mortality Rates in Males with Breast Cancer by Exposure to Finasteride | Up to 14 years
Stage 2 - Odds (or Likelihood) of Exposure to Finasteride in Male Breast Cancer Cases Relative to Controls | Up to 19 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meijer M, Thygesen LC, Green A, Emneus M, Brasso K, Iversen P, Pukkala E, Bolin K, Stavem K, Ersboll AK. Finasteride treatment and male breast cancer: a register-based cohort study in four Nordic countries. Cancer Med. 2018 Jan;7(1):254-260. doi: 10.1002/cam4.1273. Epub 2017 Dec 13. PMID 29239131